CLINICAL TRIAL: NCT01483274
Title: Pharmacologic Upregulation of Cancer Testis Antigens Followed by Vaccine Therapy for Patients With Relapsed Acute Myelogenous Leukemia (AML) Following Allogeneic Stem Cell Transplantation
Brief Title: Decitabine and Vaccine Therapy for Patients With Relapsed AML Following Allogeneic Stem Cell Transplantation
Acronym: AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Adult patient population barriers.
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13.0376
Record Dates: First submitted 2011-11-03; First posted 2011-12-01 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML; vaccine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Safety (Experimental): Decitabine and donor lymphocyte infused dendritic cell (DC).
  Interventions: Biological: Vaccine
- Vaccine (Active Comparator): Decitabine and Dendritic cell (DC) pulsed with MAGE-A1, MAGE-A3, NY-ESO-1 Peptides
  Interventions: Biological: Vaccine

INTERVENTIONS:
Biological: Vaccine — Decitabine followed by donor lymphocyte infusing and Dendritic cells pulsed with MAGE-A1, MAGE-A3, and NEY-ESO-1 vaccine
  Other Names: DAC; Dendritic cells vaccine

SUMMARY:
Patients with Acute Myelogenous Leukemia (AML) who relapse after an allogeneic stem cell transplant cell receive decitabine to up regulate cancer antigen expression, followed by a donor lymphocyte infusion and an autologous dendritic cell (DC). Vaccine Dendritic cells are pulsed with overlapping peptides derived from MAGE-A1, MAGE-A3, and NY-ESO-1.

DETAILED DESCRIPTION:
For vaccine production, mature DC will be pulsed with overlapping peptides mixes derived from full-length NY-ESO-1, MAGE-A1, and MAGE-A3.

ELIGIBILITY:
Inclusion Criteria for study enrollment:

* Signed informed consent after discussion of alternative therapies.
* The first six patients be18 to 65 years old. Patients # 7-10 will range in age from 2 - 65 years.
* Histologically or cytogenetically confirmed diagnosis of acute myelogenous leukemia prior to allogeneic SCT, with the following risk factors:

  * > second complete response, or in relapse, at the time of transplant
  * monosomy 5 or 7
  * the presence of a high FLT3/ITD allelic ratio
  * patients with detectable minimal residual disease (MRD) post-transplant
  * < 0.5% positive for recipient leukemia cells by flow cytometry

Inclusion criteria to begin study therapy:

* Patient is at least three months post-transplant.
* Patients must be off systemic immunosuppression for at least two weeks prior to the start of therapy on the study.
* ECOG performance status 0-2, Lansky performance status >70 (see Appendix 1).
* Hematologic Function: ANC: ≥ 500; Platelet count: ≥ 75.
* Renal Function:

  * Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 OR a serum creatinine based on age/gender using the Schwartz formula:
* Cardiac Function: Patient must have normal cardiac function documented within two weeks before starting of a treatment cycle 1 by:

  * Ejection fraction (> 55%) documented by echocardiogram or fractional shortening (≥ 28%) documented by echocardiogram.
* Liver Function: Total bilirubin ≤ 1.5 x normal for age, and ALT (SGPT) and AST (SGOT) ≤ 3 x normal for age.
* Room air pulse oximetry > 94%.
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of enrollment.
* Male and female patients must agree to use a medically acceptable barrier and/or chemical contraceptive method during the study and for a minimum of 3 months after the last dose of chemotherapy on this study.
* Subjects must be > 3 months and < 12 months post-SCT at the time of the first vaccination.
* Donor chimerism must be > 90%, assist at least two weeks prior to beginning treatment
* Subjects must be at least 30 days post-transplant to enroll on the study and to undergo apheresis, and must be at least three months post-transplant to begin therapy with DAC/vaccine.
* Stem cell donor source may be related or unrelated donor cord blood, related or unrelated donor bone marrow, and related or unrelated donor peripheral blood stem cell product. Donors may be no more than two HLA (A, B, C, DR, DQ) antigen mismatched with the recipient.

Exclusion Criteria:

* Patient has a history of autoimmune disease, specifically inflammatory bowel disease, systemic lupus erythematosis, or rheumatoid arthritis.
* Patient has a known systemic hypersensitivity to DAC, imiquimod, or any vaccine component.
* Patient has evidence of recurrent leukemia.
* Patient is receiving systemic corticosteroids or other immunosuppression.
* Persistent clinically significant toxicity from prior anticancer therapy that is > Grade 2 (NCI CTCAE v3.0).
* Pregnant or lactating females are excluded.
* Other active systemic malignancy other than leukemia expected to require therapy within 4 months.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Any condition which, in the opinion of the investigator, would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients with a positive result for any of the following diagnostic tests: Hep B Ag, Hep B Core Ab, Hep C Ab, HIV-1 Ab, HIV-2 Ab, HTLV-1 Ab, HTLV-2 Ab, RPR.
* Received any investigational new drug within 30 days prior to the first dose of vaccine , or are scheduled to receive an investigational new during the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Tolerance of study treatment | 4 years
  Tolerance to DAC, at least 50% dosing, and 3 of the 4 planned vaccinations during the first two cycles

SECONDARY OUTCOMES:
Disease Response | 4 years
  Assessment of Bone Marrow aspiration to check for complete or partial remission, stable disease, and disease progression by bone marrow draws at week 6 and week 12.
Immune Response | 4 years
  Assessment of post-vaccination T cell responses to MAGE-A1, MAGE-A3, and NY-ESO-1 by immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Lucas, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States